CLINICAL TRIAL: NCT04922242
Title: Assessing the Efficacy and Validity of the Welch Emotional Connection Screen (WECS) in the NICU
Brief Title: Welch Emotional Connection Screen (WECS) in the NICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Einhorn Collaborative (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAT5743
Record Dates: First submitted 2021-05-28; First posted 2021-06-10 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Premature Birth; Obstetric Labor, Premature
Keywords: nursing education; emotional connection
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — Intensive Care Units, Neonatal

STUDY DESIGN:
Intervention Model Description: Cross-sectional model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Population 1: NICU Study Staff (Experimental): Interdisciplinary Professional Clinical Staff who are employed to work as a nurse, therapist, social worker or physician in the NICU.
  Interventions: Other: NICU WECS Training
- Population 2: Mother-infant dyads in NICU (Experimental): Parent and infant dyads admitted to a NICU for over 72 hours.
  Interventions: Behavioral: Welch Emotional Connection Screen for Neonatal Intensive Care Unit

INTERVENTIONS:
Behavioral: Welch Emotional Connection Screen for Neonatal Intensive Care Unit — The Welch Emotional Connection Screen (WECS) is an investigational developmental screening tool, developed to rate the quality of the emotional connection that formed between mother and child. The screen is administered in 2-3 minutes by observing a mother and child interact, and requires the rater to critically assess 4 sub-domains of emotional connection. The NICU WECS is a clinical tool adapted for use with neonates in the NICU. Reliability of NICU staff WECS scoring will be calculated via intra-class correlations with key scores. The WECS is scored on intervals of 0.5, with a minimum of 1 (rarely--low level of connection) and maximum of 3 (mostly--high connection). Scores are used to determine the level of need for intervention.
  Arms: Population 2: Mother-infant dyads in NICU
Other: NICU WECS Training — WECS Training is an educational module consisting of an introduction of the concepts of emotional connection and autonomic co-regulation as studied by The Nurture Science Program, as well as an illustration of how these experiential constructs differ from traditional care plans that focus on educating parents to encourage "bonding" as opposed to autonomic emotional connection within the NICU. An introduction to the domains of the WECS screen as well as illustrations of these domains through video will augment the training designed for NICU staff.
  Arms: Population 1: NICU Study Staff

SUMMARY:
The purpose of this study is to assess knowledge about emotional connection, attitude about relational health, and efficacy of Welch Emotional Connection Screen (WECS) training in the NICU. The investigators seek to discern if through this didactic training, frontline NICU clinicians can be taught to reliably use the WECS to rate parent-child relational health. Additionally, the investigators seek to learn if there is construct and theoretical validity of the hospitalized infant preterm WECS by correlating WECS scores to physiological, behavioral and mental health markers for parent and infant.

DETAILED DESCRIPTION:
The Welch Emotional Connection Screen (WECS) is an investigational developmental screening tool that was developed to rate the quality of the emotional connection that formed between mother and child. When administered at 4 months of age, the scale has predictive value in determining which children will show higher risk for developmental problems at 18 months of age. The scale is administered in 2-3 minutes by observing a brief interaction between mother and child and requires the rater to critically assess 4 domains of emotional connection.

The present study will introduce an educational module for teaching NICU clinicians to critically observe mother-child interactions through use of a standardized didactic experience and structured use of the brief clinical screening tool, the WECS, and the theories around nurturing and emotional connection. In one module training session, participants will view a pre-recorded webinar on the WECS developed by the Nurture Science Program at Columbia University. During the second part of the training, participants will view and rate a set of pre-recorded parent-child interactions using the WECS. Clinicians will complete a survey and participate in a focus group discussion about their experiences with the training process and utility of the WECS in clinical practice. Determining if the WECS can be used easily and reliably by NICU clinicians will help to create new strategies that better meet the needs of all professionals involved in NICU care, as well as the families they serve.

ELIGIBILITY:
Inclusion Criteria:

* Population 1: Consenting Interdisciplinary Professional Clinical Staff who are employed to work in the NICU as a:

  * Nurse
  * Therapist
  * Social worker
  * Physician
* Population 2: Consenting parents and infants whose parents give consent by guardianship and whose physicians approve inclusion in the study.

Exclusion Criteria:

* Both populations: Refusal to consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2021-04-17 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Acceptance rate of NICU WECS and WECS Training: Focus Group | Up to 6 months
  Assess staff opinions of NICU WECS using focus groups. Responses will be coded utilizing a grounded theory hypothesis to find thematic evidence to assess the feasibility, utility, acceptability, and efficacy of the WECS in clinical practice.
Acceptance rate of NICU WECS and WECS Training: Staff Survey | Up to 6 months
  Assess staff opinions of NICU WECS using a survey. Responses will be coded utilizing a grounded theory hypothesis to find thematic evidence to assess the feasibility, utility, acceptability, and efficacy of the WECS in clinical practice.

SECONDARY OUTCOMES:
Intra-Class Correlations of Welch Emotional Connection Screen (WECS) NICU Scores | Up to 6 months
  Reliability of NICU staff WECS scoring will be calculated via intra-class correlations with key scores during training, and clinically coded WECS scores will be correlated with scores generated by a Nurture Science Program staff member. The WECS is scored on intervals of 0.5, with a minimum of 1 (rarely--low level of connection) and maximum of 3 (mostly--high connection). Scores are used to determine the level of need for intervention.
Correlation of WECS scores with Edinburgh Postnatal Depression Scale Score | Near discharge (up to 40 weeks)
  The Edinburgh Postnatal Depression Scale is a 10-item questionnaire that was developed to identify women who have postpartum depression. Items of the scale correspond to various clinical depression symptoms, such as guilt feeling, sleep disturbance, low energy, anhedonia, and suicidal ideation. Overall assessment is done by total score, which is determined by adding together the scores for each of the 10 items. Higher scores indicate more depressive symptoms.
Correlation of WECS scores with STAI Score | Near discharge (up to 40 weeks)
  The State-Trait Anxiety Inventory (Spielberger et al, 1983) comprises 2 separate self-report scales of 20 items each that measure state and trait anxiety.
Correlation of WECS scores with CES-D | Near discharge (up to 40 weeks)
  The CES-D is a 20 item self-report inventory designed to assess current but nonspecific distress rather than clinically diagnosed depression (Radloff 1977). It is the most frequently used measure in the field of infant research and maternal depression. Items probe for depressive symptoms and attitudes within the past week. Criteria are based on DSM-IV criteria for depressive disorders. A score of 16+ is traditionally used to select a depressed group. A more stringent cut-off for depression is 23+. Consistent with previous literature we will examine a low-scoring group CES-D = 0, 1, who endorse no distress.
Parent Stressor Scale (PSS): Neonatal Intensive Care Unit (NICU) | Near discharge (up to 40 weeks)
  The PSS: NICU is a 26-item self-report measure of stress assessing three dimensions of parental experience during NICU stay: Sight and Sounds, Infant Behavior and Appearance, Parental Role Alteration. Parents are asked to rate each item on a five-point Likert scale from 'not stressful' to extremely stressful'

OTHER OUTCOMES:
Correlation of WECS scores with LOS | Up to 1 year
  Correlate NICU WECS scores with quality indicators including LOS.
Correlation of WECS scores with Days on Respiratory Support | Up to 1 year
  Correlate NICU WECS scores with quality indicators including days on respiratory support.
Correlation of WECS scores with Days to Full Feeds | Up to one year
  Correlate NICU WECS scores with quality indicators including Days to full feeds.
Correlation of WECS scores with Breastfeeding Data | Up to 1 year
  Correlate NICU WECS scores with quality indicators including breastfeeding data.

CONTACTS AND LOCATIONS:
Overall Officials: Martha G. Welch, MD, Principal Investigator — Professor of Psychiatry
Locations (1):
- The Valley Hospital, Ridgewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No